CLINICAL TRIAL: NCT02339103
Title: Study of Heat and Intravenous Fluids for Exogenous Rewarming (SHIVER)
Brief Title: Study of Heat and Intravenous Fluids for Exogenous Rewarming
Acronym: SHIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 31036
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Hypothermia
Keywords: arteriovenous anastomoses; accidental hypothermia; rewarming
MeSH Terms: conditions — Hypothermia; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shivering only (No Intervention): Pt placed in sleeping bag and warmed by shivering only
- Warmed IV fluids (Experimental): 2 Liter of 42 degree celsius normal saline
  Interventions: Other: Warmed IV fluids
- Warmed perfusion pads (Experimental): Warmed perfusion pads placed to palms and soles to rewarm through arteriovenous anastomoses
  Interventions: Other: Warmed perfusion pads

INTERVENTIONS:
Other: Warmed IV fluids — 1 Liter of warmed IV fluids at 42 degrees celsius
  Arms: Warmed IV fluids
Other: Warmed perfusion pads — Neoprene perfusion pads placed on the palms and soles to rewarm through focusing on the arteriovenous anastomoses
  Arms: Warmed perfusion pads

SUMMARY:
The purpose of this study is to compare two novel active rewarming techniques in mildly hypothermic people. Volunteers will undergo 3 cooling trials in a circulating bath at 14 degrees celsius and will then be rewarmed with either shivering alone, warmed iv fluids (IVF), or water perfusion pads applied to the hands and feet. The investigators hypothesize that both heated IVF and water perfusion pads to the arteriovenous anastomoses (AVAs) will prove to provide significantly superior rewarming rates than shivering alone.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy male or female over 18 years of age

Exclusion Criteria:

* No heart/blood pressure/cholesterol medications.
* No history of Raynaud's disease or any other condition (including asthma) that could be aggravated by cold-water immersion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Rate of rewarming | 60 minutes
  Track to rate of rewarming of each arm

REFERENCES:
- [Result] Christensen ML, Lipman GS, Grahn DA, Shea KM, Einhorn J, Heller HC. A Novel Cooling Method and Comparison of Active Rewarming of Mildly Hypothermic Subjects. Wilderness Environ Med. 2017 Jun;28(2):108-115. doi: 10.1016/j.wem.2017.02.009. Epub 2017 May 12. PMID 28506514